CLINICAL TRIAL: NCT03653923
Title: Neurophysiological Correlates of Exposition Therapy in Spider Phobia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 481/2018BO2
Record Dates: First submitted 2018-07-24; First posted 2018-08-31 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-07

CONDITIONS: Phobic Disorders
MeSH Terms: conditions — Phobic Disorders | interventions — Implosive Therapy; Psychotherapy

STUDY DESIGN:
Intervention Model Description: Waiting-List RCT with crossover after Treatment (Waiting-List will be treated, treated subjects will rest)
Masking Description: Psychotherapeutic Investigation - No masking possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Waiting-List (Experimental)
  Interventions: Behavioral: Exposure Therapy
- Treatment (Experimental)
  Interventions: Behavioral: Exposure Therapy
- Healthy Controls (No Intervention): Not randomized healthy control group for comparison to normal functioning

INTERVENTIONS:
Behavioral: Exposure Therapy — Before the treatment, subjects will have one session of psychoeducation in which the rationale for the treatment is explained. In each therapy session subjects are exposed to 20 trials (each lasting 40s) of guided exposure by a psychotherapist. Further, 20 control trials of equal length are assessed in which subjects work with an earthworm. Each session lasts for approximately 90 minutes. During the therapy additional anxiety coping strategies (e.g., controlled breathing, attention refocusing, cognitive reappraisal) are trained.
  Subjects of the waiting-list will be treated in the second study phase.
  Other Names: Psychotherapy
  Arms: Treatment; Waiting-List

SUMMARY:
This study aims to investigate the neurophysiological correlates of spider phobia and its treatment with CBT based Exposure Therapy. This is the first study to investigate the neurophysiological correlates of Exposure Therapy in situ by means of functional Near-Infrared Spectroscopy (fNIRS).

30 spider phobic patients will be assessed and randomly allocated to 5 sessions of exposure therapy or waiting-list. Further, 30 non-phobic control subjects will be assessed (primary assessment only).

During Exposure Therapy, changes in blood oxygenation will be measured with fNIRS in areas of the Cognitive Control Network. Regions of interest are the bilateral dorsolateral prefrontal cortex (DLPFC), bilateral inferior frontal gyrus (IFG) and somatosensory association cortex (SAC). Before the treatment, subjects will have one session of psychoeducation in which the rationale for the treatment is explained. In each therapy session subjects are exposed to 20 trials (each lasting 40s) of guided exposure by a psychotherapist. Further, 20 control trials of equal length are assessed in which subjects work with an earthworm. During the therapy additional anxiety coping strategies (e.g., controlled breathing, attention refocusing, cognitive reappraisal) are trained. After the treatment or waiting-list phase, treatment conditions are switched: The waiting list will be treated and the treated subject will wait for approximately 6 weeks.

Before treatment (primary assessment), after treatment (secondary assessment) and after study completion (final assessment), additional combined NIRS EEG measurements are done. On a peripheral physiological level heart rate and EMG of the facial corrugator supercilii are measured. During these measurements subjects are asked to watch 10s lasting video clips showing spiders (experimental condition) or pets (dogs and cats). On a psychometric level, spider phobia will be assessed by questionnaires (SPQ, FSQ, SBQ) and behavioral assessments.

ELIGIBILITY:
Inclusion Criteria:

* Spider Phobia or no fear of spiders
* Age between 18 and 50
* normal vision (or corrected with glasses)
* German mother tongue or comparable knowledge

Exclusion Criteria:

* pregnancy
* medication with exception of contraceptive medication
* acute or chronic disease that affects brain functioning (other mental diagnosis than spider phobia, cardial diseases, diabetes, kidney diseases, concussion)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
fNIRS | Before Treatment (Primary Assessment, approximately week 1), after treatment completion (secondary assessment, approximately week 6) and after study completion (final assessment, approximately week 12); During Exposure Therapy
  Oxygenated and Deoxygenated Blood in the cerebral cortex will be measured with functional Near-Infrared Spectroscopy. Analysed will be Changes in Oxygenated Blood from Pre to Post-Measurement and between Control Conditions (EarthWorm) and Experimental Conditions (Working with Spiders). At Pre-Testing, the clinical population will be compared to the healthy controls.

SECONDARY OUTCOMES:
spider phobia questionnaire | Before Treatment (Primary Assessment, approximately week 1), after treatment completion (secondary assessment, approximately week 6) and after study completion (final assessment, approximately week 12)
  Range SPQ: 0 to 31, high values indicate high fear of spiders
Behavioral Measures | Before Treatment (Primary Assessment, approximately week 1), after treatment completion (secondary assessment, approximately week 6) and after study completion (final assessment, approximately week 12)
  Avoidance with respect to spiders will be assessed on a behavioral scale
  1. = Spider is 5 m away (in a jar)
  2. = Patient watches pictures of spiders while the spider is 5 m away
  3. = spider is 2 m away (in a jar)
  4. = spider is 0.5 m away (in a jar)
  5. = spider is directly in front of the subject (in a jar)
  6. = spider is taken out of the jar into a larger tub
  7. = patient touches the spider with a pen
  8. = the spider is on the (covered) hand of the patient
  9. = patient touches the spider with his finger
  10. = spider walks on the hand of the patient
  11. = spider walks up the arm of the patient
Peripheral Physiology | Before Treatment (Primary Assessment, approximately week 1), after treatment completion (secondary assessment, approximately week 6) and after study completion (final assessment, approximately week 12)
  Heart rate and electromyography of the facial corrugator supercilii will be assessed
EEG/EKP | Before Treatment (Primary Assessment, approximately week 1), after treatment completion (secondary assessment, approximately week 6) and after study completion (final assessment, approximately week 12)
  Event-Related Potentials will be assessed with EEG
Fear of Spiders Questionnaire | Before Treatment (Primary Assessment, approximately week 1), after treatment completion (secondary assessment, approximately week 6) and after study completion (final assessment, approximately week 12)
  Range FSQ: 18 to 126, high values indicate high fear of spiders
Spider-Phobia-Beliefs Questionnaire | Before Treatment (Primary Assessment, approximately week 1), after treatment completion (secondary assessment, approximately week 6) and after study completion (final assessment, approximately week 12)
  Range SBQ (mean): 0 to 100%, high values indicate high maladaptive beliefs of spiders
Visual analogue scales | During each exposure session (week 1 to 5) and during EEG assessments (Before Treatment (Primary Assessment, approximately week 1), after treatment completion (secondary assessment, approximately week 6) and after study completion (approximately week 12)
  During exposure fear, disgust and aviodance will be rated after each trial by the subject on a scale from 1 (not at all) to 9 (very much)

CONTACTS AND LOCATIONS:
Overall Officials: David Rosenbaum, Dipl.-Psych., Principal Investigator — Universitiy Hospital of Tuebingen
Locations (1):
- Department of Psychiatry and Psychotherapy, University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be sent after enquiry